CLINICAL TRIAL: NCT01460914
Title: Outcomes of Cutaneous T-Cell Lymphoma and Chronic Graft-Versus-Host Disease in Patients Treated With Extracorporeal Photopheresis
Brief Title: Outcomes of Cutaneous T-Cell Lymphoma and Graft-Versus-Host Disease With Extracorporeal Photopheresis Treatment
Status: Completed | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Frederick Lansigan, Assistant Professor of Medicine, Dartmouth-Hitchcock Medical Center
Other Study IDs: D11271
Record Dates: First submitted 2011-10-19; First posted 2011-10-27 (Estimated); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Cutaneous T Cell Lymphoma; Graft Versus Host Disease
Keywords: ECP; CTCL; Extracorporeal photopheresis; Cutaneous T Cell Lymphoma; GVHD; Graft versus host disease
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Graft vs Host Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Extracorporeal Photopheresis (ECP) is a form of apheresis and photodynamic therapy in which the peripheral blood is treated with 8-methoxypsoralen, which is then activated with UV light. ECP is currently a standard therapy for cutaneous T-cell lymphoma (CTCL) and is also effective for graft-versus-host disease (GVHD). The investigators would like to study the outcomes (response rates) of patients receiving ECP treatment and other factors relating to their disease and treatment, as well as procedural events, such as complications.

DETAILED DESCRIPTION:
The investigators intend to report outcomes from the inception of this procedure at Dartmouth-Hitchcock Medical Center (DHMC) in May 2008 through 9/30/11. Additionally, the investigators would like to maintain a prospective database of these patients so that new patient data can be collected for updating of outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients who receive Extracorporeal Photopheresis treatment
* Treated at Dartmouth-Hitchcock Medical Center
* Must be 18 years or older

Exclusion Criteria:

- None specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who receive ECP treatment at DHMC
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2011-10-01 (Actual); Primary Completion 2015-01-06 (Actual); Study Completion 2015-01-06 (Actual)

PRIMARY OUTCOMES:
Response rates | 1 year
  Response rates to ECP treatment

SECONDARY OUTCOMES:
Complications | 1 year
  Complications to ECP procedures

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Lansigan, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

REFERENCES:
- [Result] Weber LL, Dunbar NM, Meehan KR, Szczepiorkowski ZM, Lansigan F. Successful implementation of a rural extracorporeal photopheresis program for the treatment of cutaneous T-cell lymphoma and chronic graft-versus-host disease in a rural hospital. J Clin Apher. 2015 Dec;30(6):359-63. doi: 10.1002/jca.21382. Epub 2015 Feb 17. PMID 25691106